CLINICAL TRIAL: NCT01561924
Title: An Exploratory Non-interventional Study of Ex-vivo Spiking Followed by Thromboelastography as a Method for Predicting the Efficacy of Recombinant Activated Human FVII (rFVIIa, NovoSeven®) in Adult Congenital Haemophilia A or B Patients With Inhibitors
Brief Title: Prediction of the Efficacy of Activated Recombinant Human Factor VII in Adult Congenital Haemophilia A or B Patients With Inhibitors by Use of Thromboelastography
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: F7HAEM-1675
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ex vivo (Experimental)
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — Subjects will be called to attend the clinic in a non-bleeding state. Blood samples will be drawn for thromboelastogram profiling and will be in-vitro spiked with different doses of activatated recombinant human factor VII.
  Other Names: activated recombinant human factor VII

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to evaluate the basal and spiked TEG® (Thromboelastography) or ROTEM® (Thromboelastometry) profiles of frequently bleeding haemophilia subjects with inhibitors in a non-bleeding state.

DETAILED DESCRIPTION:
The TEG parameters are: R time (Reaction Time), K time (K Time (arbitrary measurement)), a (a angle), MA (Maximum Amplitude) and LY30 (Lysis 30 min after MA) while the ROTEM parameters are: CT (Clotting Time), CFT (Clot Formation Time), a (a angle), MCF (Maximum Clot Firmness) and LI60 (Lysis index 60 min after CT)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of congenital haemophilia A or B with a FVIII:C clot activity or FIX:C clot activity, respectively, less than 5%
* Presently use of activated recombinant human factor VII (NovoSeven®) as haemostatic agent for preventive treatment or treatment of bleeding episodes
* A documented historical or present record for the presence of inhibitors to factor VIII or IX, respectively
* A documented history of 2 or more joint bleeding episodes during the preceding 12 months
* Subjects must be in a non-bleeding state (i.e. no clinical manifestations of active bleeds)

Exclusion Criteria:

* Subjects who have received any haemostatic treatment for a bleeding episode within the last 7 days prior to this trial
* Immune tolerance therapy within the last 30 days prior to this trial
* Clinically relevant coagulation disorders other than congenital haemophilia A or B
* Thrombocytopenia (platelet count below 60,000 platelets/mcl)
* Prophylactic haemostatic treatment within 3 days prior to this trial

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-11; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
TEG parameters obtained at baseline and with activated recombinant human factor VII
ROTEM parameters obtained at baseline and with activated recombinant human factor VII

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (7):
- United States (4):
  - Novo Nordisk Investigational Site, Berkeley, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
- Novo Nordisk Investigational Site, Århus N, Denmark
- Novo Nordisk Investigational Site, Lyon, France
- Novo Nordisk Investigational Site, London, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com